CLINICAL TRIAL: NCT02067754
Title: Circulating Free DNA Analysis in Gastrointestinal Cancer, Genitourinary Cancer, Rare Cancer
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Professor, Samsung Medical Center
Other Study IDs: 2013-06-076
Record Dates: First submitted 2014-02-10; First posted 2014-02-20 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Gastric Cancer
Keywords: The mutation profiling of circulating free DNA
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — * From each enrolled patient who meets the inclusion/exclusion criteria, blood samples will be collected 10 mL blood sample will be collected at the baseline and every cycles of tumor evaluation.
  * 20 of 5µm unstained sections will be collected at the time of study entry.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- metastatic Cancer: metastatic gastrointestinal cancer, genitourinary cancer , rare cancer with treated any anti-cancer therapy

SUMMARY:
The investigators planned this study to Patients with histologically confirmed metastatic gastrointestinal cancer, genitourinary cancer , rare cancer with treated any anti-cancer therapy : Extra blood sample collection during routine blood sampling.

DETAILED DESCRIPTION:
Metastasis is a leading cause of cancer related deaths and is also one of the poorly understood aspects of cancer progression. During metastatic outgrowth, a cancer cell from a primary tumor locally invades the surrounding tissue, undergoes intravasation to enter hematogenous circulation and translocates to distant tissues through extravasation, survives and adapts to the foreign microenvironment leading to formation of a macroscopic secondary tumor (Figure 1, Chaffer and Weinberg (2011)). Several cancer therapies have been introduced in the last few decades from cytotoxics to targeted agents. However, these therapies fail to modulate growth of metastatic tumor cells which are often resistant, with most cancer patients succumbing to metastatic disease. There is a key need to further the understanding of metastatic disease in order to develop newer therapies. A central and somewhat unaddressed question is whether this acquisition of malignant traits occurs as an inevitable consequence of tumor progression or as an accidental product thereof. A widely accepted but not so well proven model of primary tumor formation suggests that cancer cells acquire a sequence of genetic and epigenetic alterations, each of which confers one or another form of increased fitness.

Figure 1: The metastatic cascade. Metastasis can be envisioned as a process that occurs in two major phases: (i) physical translocation of cancer cells from the primary tumor to a distant organ and (ii) colonization of the translocated cells within that organ. (A) To begin the metastatic cascade, cancer cells within the primary tumor acquire an invasive phenotype. (B) Cancer cells can then invade into the surrounding matrix and toward blood vessels, where they intravasate to enter the circulation, which serves as their primary means of passage to distant organs. (C) Cancer cells traveling through the circulation are Circulating free DNA. They display properties of anchorage-independent survival. (D) At the distant organ, Circulating free DNA exit the circulation and invade into the microenvironment of the foreign tissue. (E) At that foreign site, cancer cells must be able to evade the innate immune response and also survive as a single cell (or as a small cluster of cells). (F) To develop into an active macrometastatic deposit, the cancer cell must be able to adapt to the microenvironment and initiate proliferation.

It is somewhat accepted that tumors are clonally derived through unregulated growth of single cells that have likely accumulated the necessary number and types of heritable genetic and genomic alterations. Despite the monoclonal origin of cancer, the investigators see many tumors display a large amount of genetic, genomic and signaling heterogeneity. This heterogeneity is also believed to be one of the main drivers of metastasis. This heterogeneity has implications for understanding the disease progression landscape on one hand and diagnosis and treatment decisions on other. It is therefore of direct clinical importance to study the similarities and differences between the primary tumor and metastatic variants

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years
* Patients with histologically confirmed metastatic gastrointestinal cancer, genitourinary cancer , rare cancer with treated any anti-cancer therapy
* Written informed consent form

Exclusion Criteria:

* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical condition that would interfere with the subject's safety.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically confirmed cancer patients
Sampling Method: Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2013-09-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Circulating tumor cell | 1years
  To survey the mutation profiling of circulating free DNA in gastrointestinal cancer, genitourinary cancer, and rare cancer.

SECONDARY OUTCOMES:
mutation profiling of circulating free DNA | 1years
  1. To prospectively collect blood samples from patients and construct clinical database of gastrointestinal cancer, genitourinary cancer, rare cancer patients
  2. To define genotypes of circulating free DNA which will likely to response to anti-cancer therapy

OTHER OUTCOMES:
Circulating Free DNA Analysis in Gastrointestinal Cancer, Genitourinary Cancer | From date of start of chemotherapy treatment by Circulating free DNA until the date of first progression or date of death from any cause.
  The objective of this collaboration will be to evaluate the performance of next generation sequencing assay on mutation detection using matched plasma and primary tumor from various types of cancer.
  The ultimate goal is to develop an ultra sensitive assay of mutation detection for early diagnosis, monitoring disease progression and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, MD,PhD, Principal Investigator — Division of oncologyu, Department of Medicine, Samsung Medical Center
Locations (1):
- Samsung Medical center, Seoul, South Korea

REFERENCES:
- [Background] 1. Lower EE etal. Impact of metastatic ER and PR status on survival. Breast Cancers and Treat. 90. 65-75. 2005. 2. Regitnig P et al. Change of Her-2/neu status in a subset of distant metastases from breast carcibnoma. J Pathol. 203 94) 918-26, 2004. 3. Cristofanilli M. Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med 351:781-91. 4. Riethdorf S, Fritsche H, Muller V, Rau T, Schindlbeck C, Rack B, Janni W, Coith C, Beck K, Janickje F, Jackson S, Gornet T, Cristofanilli M, Pantel K. Detection of circulating tumor cells in peripheral blood of patients with metastatic breast cancer: a validation study of the CellSearch system. Clin Cancer Res 13:920-8. 2007 5. Cristofanilli M, Broglio KR, Guarneri V, Jackson S, Fritsche HA, Islam R, Dawood S, Reuben JM, Kaum SW, Lara JM, Krishnamurthy S, Ueno NT, Hortobagyi GN, Valero V. Circulating tumor cells in metastatic breast cancer: biologic staging beyond tumor burden. Clin Breast Cancer 7:471-9, 2007.
- [Derived] Kim ST, Lee WS, Lanman RB, Mortimer S, Zill OA, Kim KM, Jang KT, Kim SH, Park SH, Park JO, Park YS, Lim HY, Eltoukhy H, Kang WK, Lee WY, Kim HC, Park K, Lee J, Talasaz A. Prospective blinded study of somatic mutation detection in cell-free DNA utilizing a targeted 54-gene next generation sequencing panel in metastatic solid tumor patients. Oncotarget. 2015 Nov 24;6(37):40360-9. doi: 10.18632/oncotarget.5465. PMID 26452027